CLINICAL TRIAL: NCT00044759
Title: A Randomized, Open-Label, Multi-Center, Comparative Study of the Efficacy and Safety of Piperacillin/Tazobactam to Cefepime for the Empiric Treatment of Neutropenic Fever in Patients With a Hematologic Malignancy or Lymphoma
Brief Title: Study Comparing the Safety and Efficacy of Piperacillin/Tazobactam to Cefepime in Patients With Hematologic Malignancy or Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Purpose: Treatment
Other Study IDs: 0910B1-308
Record Dates: First submitted 2002-09-04; First posted 2002-09-06 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: Hematologic Neoplasms
Keywords: Hematologic; Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms | interventions — Piperacillin; Tazobactam; Piperacillin, Tazobactam Drug Combination

INTERVENTIONS:
Drug: Piperacillin/Tazobactam (Tazocin)

SUMMARY:
To compare the safety and efficacy of piperacillin/tazobactam (4 g/500 mg) administered intravenously every 6 hours to cefepime (2 g) administered intravenously every 8 hours for the empiric treatment of neutropenic fever in patients with a hematologic malignancy or lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized male and female patients, 18 years of age or older
* Patients who have leukemia (acute lymphocytic leukemia [ALL], acute myelogenous leukemia [AML], chronic lymphocytic leukemia [CLL], chronic myelogenous leukemia [CML]), that is newly diagnosed, who have had initial induction, re-induction, or intensification chemotherapy or who have had a bone marrow (allogenic, syngeneic, or autologous) or peripheral blood stem-cell transplant OR Patients with lymphoma, Hodgkin's disease, multiple myeloma, myelodysplastic syndrome or myelodysplasia (refractory anemia [RA], refractory anemia with ringed sideroblasts [RARS], refractory anemia with excess blasts [RAEB], refractory anemia with excess blasts in transformation to leukemia [RAEB-T], or chronic myelomonocytic leukemia [CMML].
* Fever, defined as an oral temperature of ≥ 37.9°C /100.2°F, a rectal temperature ≥ 38.4°C /101.4°F, or a tympanic temperature ≥ 38°C /100.4°F

Exclusion Criteria:

* The presence of any clinically acute or chronic disease or condition that, in the opinion of the investigator, may interfere with the patient's ability to safely comply with the conditions of the protocol, or could preclude the evaluation of the patient's response or could make the completion of the therapy unlikely
* Neutropenia associated with syndromes that are not associated with a high risk of bacterial infection (eg. chronic benign neutropenia or Kostmann's syndrome)
* Neutropenia due to primary bone marrow failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (33):
- United States (28):
  - Little Rock, Arkansas
  - Los Angeles, California
  - Denver, Colorado
  - Gainesville, Florida
  - North Miami, Florida
  - Ocala, Florida
  - St. Petersburg, Florida
  - Thomasville, Georgia
  - Chicago, Illinois
  - Iowa City, Iowa
  - Louisville, Kentucky
  - Camden, New Jersey
  - Hackensack, New Jersey
  - Buffalo, New York
  - New York, New York
  - Rochester, New York
  - The Bronx, New York
  - Valhalla, New York
  - Tulsa, Oklahoma
  - Philadelphia, Pennsylvania
  - Sayre, Pennsylvania
  - Upland, Pennsylvania
  - West Reading, Pennsylvania
  - Providence, Rhode Island
  - Columbia, South Carolina
  - Houston, Texas
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Canada (5):
  - Hamilton
  - Montreal
  - Ottawa
  - Saskatoon
  - Winnepeg